CLINICAL TRIAL: NCT07293806
Title: Study Protocol for a Randomised Controlled Trial of Dance-movement Therapy for Adolescents With Depression
Brief Title: Dance-movement Therapy in the Treatment of Adolescent Depression
Acronym: DMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Finnish Medical Foundation (Network); Finnish Institute for Health and Welfare (Other Government); University of Helsinki (Other)
Responsible Party: Principal Investigator, Riikka Valjakka, Medical doctor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/391/2021
Record Dates: First submitted 2022-08-29; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: adolescents; depression; therapy; dance; movement
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Dance movement therapy group intervention (DMT) is compared with treatment as usual (TAU)
Masking Description: It is not possible to mask participants or care providers. No need for masking of investigator, since the primary outcome measures are self-reporting questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance movement therapy (Experimental): A group of 5-6 patients is recieving Dance movement group therapy once a week for 12 weeks
  Interventions: Other: Dance movement therapy
- Treatment as usual (No Intervention): Treatment as usual in youth psychiatric outpatient clinic

INTERVENTIONS:
Other: Dance movement therapy — A group therapy model for treatment of depression by dance movement therapist. Study consist of 12 therapy sessions, each session lasting 1hour 15minutes. There will be 6 patients in each group.
  Arms: Dance movement therapy

SUMMARY:
The aim of this research is to measure the effectiveness of Dance movement therapy in the treatment of adolescent depression.

DETAILED DESCRIPTION:
Research will start by recruitment of 140 patients (aged 13-17 years) from youth psychiatric outpatient clinic in Helsinki University Central hospital. They will be randomized to two groups. The intervention group will attend Dance movement therapy (DMT) for 12 weeks and the control group is getting treatment as usual (TAU). The outcome will be measured with self-report questionnaires and interviews measuring symptoms of depression and body image. Outcome measurements will be done before intervention, after intervention and 3 months after intervention has finished. The research will start in September 2022 and continue until the end of 2027. The results will be published in medical scientific journals during the year 2027

.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of medium or severe depression; BDI 16 points or more. At least 4/9 symptoms of depression in K-SADS-PL interview

Exclusion Criteria:

* Acute psychosis, psychotic depression, personality disorder, severe anorexia, substance misuse that is on a critical level

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-21) | baseline, 8 weeks, 12 weeks, 6 months
  The self-report questionnaire to assess depressive symptoms, minimum 0 points, maximum 63 points, more severe depression with higher scores
Young Person's Clinical Outcomes in Routine Evaluation (YP-Core) | baseline, 8 weeks, 12 weeks, 6 months
  The self- report questionnaire to measure depressive and overal symptoms in youth, minimum 0 points, maximum 40 points, or median of scores, higher scores indicating more symptoms

SECONDARY OUTCOMES:
Adolescent Depression Rating Scale (ADRS) | baseline, 12 weeks, 6 months
  Clinical interview to measure depressive symptoms in youth, minimum 0 and maximum 60 points, highers scores indicating more severe depression
Body Image assessment | baseline, 12 weeks, 6 months
  Self-report questionnaire to assess body image/experience, 11 items with minimum 11 and maxomum 77 points, a qualitative scale

CONTACTS AND LOCATIONS:
Overall Officials: Mauri Marttunen, Prof emer, Study Chair — University of Helsinki; Henna Haravuori, Docent, Study Director — Finnish Institue for Health and Welfare
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Adolecent mental health services, Helsinki, Helsinki

IPD SHARING:
Plan to Share IPD: No
Individual deidentified participant data will not be shared due to legal and ethical restrictions and institute policy; other documents will be available (e.g., study protocol, statistical analysis plan, etc.); data (means, distributions etc.) for meta-analyses and like will be provided, data will be available earliest 2027 and according to study's institutional permissions; for researchers in esteemed institutes, with safe digital methods.

REFERENCES:
- [Background] Hyvonen K, Pylvanainen P, Muotka J, Lappalainen R. The Effects of Dance Movement Therapy in the Treatment of Depression: A Multicenter, Randomized Controlled Trial in Finland. Front Psychol. 2020 Aug 12;11:1687. doi: 10.3389/fpsyg.2020.01687. eCollection 2020. PMID 32903394
- [Background] Cooney GM, Dwan K, Greig CA, Lawlor DA, Rimer J, Waugh FR, McMurdo M, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD004366. doi: 10.1002/14651858.CD004366.pub6. PMID 24026850
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Jeong YJ, Hong SC, Lee MS, Park MC, Kim YK, Suh CM. Dance movement therapy improves emotional responses and modulates neurohormones in adolescents with mild depression. Int J Neurosci. 2005 Dec;115(12):1711-20. doi: 10.1080/00207450590958574. PMID 16287635
- [Background] Karkou V, Aithal S, Zubala A, Meekums B. Effectiveness of Dance Movement Therapy in the Treatment of Adults With Depression: A Systematic Review With Meta-Analyses. Front Psychol. 2019 May 3;10:936. doi: 10.3389/fpsyg.2019.00936. eCollection 2019. PMID 31130889
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Koch SC, Riege RFF, Tisborn K, Biondo J, Martin L, Beelmann A. Effects of Dance Movement Therapy and Dance on Health-Related Psychological Outcomes. A Meta-Analysis Update. Front Psychol. 2019 Aug 20;10:1806. doi: 10.3389/fpsyg.2019.01806. eCollection 2019. PMID 31481910
- [Background] Millman LSM, Terhune DB, Hunter ECM, Orgs G. Towards a neurocognitive approach to dance movement therapy for mental health: A systematic review. Clin Psychol Psychother. 2021 Jan;28(1):24-38. doi: 10.1002/cpp.2490. Epub 2020 Jul 8. PMID 32539160
- [Background] Radovic S, Gordon MS, Melvin GA. Should we recommend exercise to adolescents with depressive symptoms? A meta-analysis. J Paediatr Child Health. 2017 Mar;53(3):214-220. doi: 10.1111/jpc.13426. Epub 2017 Jan 10. PMID 28070942
- [Background] Rohricht F, Papadopoulos N, Priebe S. An exploratory randomized controlled trial of body psychotherapy for patients with chronic depression. J Affect Disord. 2013 Oct;151(1):85-91. doi: 10.1016/j.jad.2013.05.056. Epub 2013 Jun 14. PMID 23769289
- [Background] Gergov V, Lahti J, Marttunen M, Lipsanen J, Evans C, Ranta K, Laitila A, Lindberg N. Psychometric properties of the Finnish version of the Young Person's Clinical Outcomes in Routine Evaluation (YP-CORE) questionnaire. Nord J Psychiatry. 2017 May;71(4):250-255. doi: 10.1080/08039488.2016.1270352. Epub 2017 Jan 13. PMID 28084134
- [Background] Revah-Levy A, Birmaher B, Gasquet I, Falissard B. The Adolescent Depression Rating Scale (ADRS): a validation study. BMC Psychiatry. 2007 Jan 12;7:2. doi: 10.1186/1471-244X-7-2. PMID 17222346

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT07293806/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT07293806/ICF_001.pdf